CLINICAL TRIAL: NCT00683579
Title: Neurocognitive Assessment in Youth Initiating HAART
Status: Completed | Type: Observational
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Other Study IDs: ATN 071
Record Dates: First submitted 2008-05-21; First posted 2008-05-23 (Estimated); Last update posted 2017-02-28 (Actual); Status verified 2016-02

CONDITIONS: HIV Infections
Keywords: HAART; DHHS guidelines; Treatment Naive
MeSH Terms: conditions — HIV Infections | interventions — Antiretroviral Therapy, Highly Active

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (4):
- 1: Participants with CD4+ T cells above 350 cells/mm3 and HIV RNA >1,000 copies/ml who are initiating HAART with possibility of de-intensification (early treatment).
  Interventions: Drug: Early Treatment with HAART
- 2: Participants with CD4+ T cells above 350 cells/mm3 and HIV RNA >1,000 copies/ml who are not initiating treatment.
  Interventions: Other: No treatment
- 3: Participants with CD4+ T cells < 350 cells/mm3 who are initiating treatment.
  Interventions: Drug: HAART Treatment - standard care
- 4: Participants with CD4+ T cells < 350 cells/mm3 who are not initiating treatment.
  Interventions: Other: No treatment

INTERVENTIONS:
Drug: Early Treatment with HAART — HAART with possibility of de-intensification
  Groups: 1
Other: No treatment — No treatment. For group 2, participants do not yet meet DHHS guidelines. For group 4, treatment is not initiated due to unwillingness or providers' expectation of poor adherence.
  Groups: 2; 4
Drug: HAART Treatment - standard care — Initiation of HAART per DHHS guidelines, i.e. starting treatment and CD4+ T cells less than 350 cells/mm3 or HIV RNA >100,000 copies/ml
  Groups: 3

SUMMARY:
ATN 071 is a prospective cohort study comparing neurocognitive functioning in four groups of youth, age 18-24: Two groups with CD4+ T cells above 350 cells/mm3 and HIV RNA >1,000 copies/ml, one initiating HAART (Group 1) and the other not initiating treatment (Group 2); and two groups with CD4+ T cells < 350 cells/mm3, one initiating treatment (Group 3) and the other not initiating treatment (Group 4). Groups 2 and 3 represent standard of care. Group 1 and a portion of group 2 will be co-enrolled in ATN 061 and will be randomly assigned to group by that protocol.

ELIGIBILITY:
Inclusion Criteria:

Groups 1 and 2 (If co-enrolling in ATN 061)

* HIV positive participants age 18 years and 0 days to 24 years and 364 days (the lower age limit of this study is driven by the restriction of ATZ use to age 18 and greater);
* Groups 1 and 2: CD4+ T cells above 350 cells/mm3 and HIV RNA >1,000 copies/ml, as determined by two consecutive measures within 6 months of entry with the second measure being collected at pre-entry to ATN 061;
* Infected with HIV after the age of nine via behavioral means;
* Naïve to ART except for HAART for PMTCT for six months or less with at least six months since the time of exposure;
* HIV genotype without major resistance mutations to the recommended ATV-r based HAART regimens;
* Able to provide written informed consent as determined by local Institutional Review Boards;
* Fluent in English or Spanish.

Group 2, enrolled in ATN 071 and not ATN 061

* CD4+ T cells above 350 cells/mm3 and HIV RNA >1,000 copies/ml, as determined by most recent laboratory evaluations available within 4 months prior to entry;
* Not prescribed HAART according to DHHS guidelines.

Groups 3 and 4:

* HIV positive participants age 18 years and 0 days to 24 years and 364 days;
* Infected with HIV after the of age nine via behavioral means;
* Naïve to ART except for HAART for PMTCT for six months or less with at least six months since the time of exposure;
* Able to provide written informed consent as determined by local Institutional Review Boards;
* Fluent in English or Spanish.
* CD4+ T cells < 350 cells/mm3, as determined by most recent laboratory evaluations available within 4 months prior to entry.

Group 3 ONLY:

* Participant initiating HAART.

Group 4 ONLY:

* HAART has not been prescribed due to either participant's refusal to initiate HAART or provider's concerns about participant's predicted inability to adhere to regimen.

Exclusion Criteria:

Groups 1 and 2:

* For Groups 1 and 2: any history of an AIDS-defining illness;
* Active drug or alcohol use or dependence that, in the opinion of the site personnel, would interfere with meeting study requirements;
* History of cognitive or motor impairment due to non-HIV-related conditions (for example, prematurity, cerebral palsy, closed head injury, CNS cancer or cranial irradiation, etc.) or psychosis. Youth with diagnoses of learning disabilities or attention deficit hyperactivity disorder will be allowed in the study;
* Enrollment of youth with chronic or acute medical conditions other than HIV that could potentially impact upon neurocognitive functioning requires protocol chair approval.
* Pregnancy at any time during the study including entry.

Ages: 18 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: English or Spanish speaking youth, 18 years 0 days to 24 years 364 days, with HIV-1 infection acquired after age 9 via behavioral means, in the following immunological and treatment categories:
  1. Early initiation of HAART and enrolled in 061 Arm A; CD4+ T cells above 350 cells/mm3 and HIV RNA >1,000 copies/ml;
  2. Initiation of HAART per DHHS guidelines (standard of care) but not yet meeting criteria. There will be 25 participants from ATN 061 preferentially enrolled into this protocol; an additional 25 participants will be enrolled with similar biomedical characteristics.
  3. Initiation of HAART per DHHS guidelines (not part of ATN 061).
  4. Meeting DHHS guidelines for initiating HAART, but not initiating due to unwillingness or providers' expectation of poor adherence.
Sampling Method: Non-Probability Sample
Enrollment: 220 (Actual)
Dates: Start 2007-12; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
The impact of early initiation of HAART on preventing neurocognitive decline in HIV infected adolescents compared to no treatment and initiation following current guidelines. | 3 years

SECONDARY OUTCOMES:
Assess youth who meet current DHHS guidelines for initiating HAART but either refuse to start HAART or are not prescribed HAART because of concerns about adherence. | Baseline assessment (not longitudinal)
To assess if de-intensification of HAART as will occur in Arm A of ATN 061 can minimally maintain neurocognitive gains made with one year of HAART. | 3 years
To assess the relationship of neurocognitive functioning to CD4+ and viral load at baseline in adolescents with HIV-1 infection (groups 1 and 2 versus 3 and 4). | 3 years
To correlate neurocognitive change with changes in CD4+ and viral loads within groups. | 3 years
To assess the incidence of HIV-associated dementia and minor cognitive-motor disorder in adolescents with risk-acquired HIV infection. | 3 years
To evaluate the relationship of current substance abuse to neurocognitive deficits in youth with risk-acquired HIV. | 3 years
To assess the relationship of neurocognitive functioning to available biomarkers within the subset of participants co-enrolled in ATN 061 (for example, immune activation markers, viral phenotype, CD4 and CD8 subsets). | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Sharon Nichols, Study Chair — Adolescent Trials Network
Locations (21):
- United States (20):
  - Children's Hopsital of Los Angeles, Los Angeles, California
  - University of Southern California - IMPAACT Site, Los Angeles, California
  - University of California at San Francisco, San Francisco, California
  - Children's Hospital of Denver - IMPAACT Site, Aurora, Colorado
  - Childrens National Medical Center, Washington D.C., District of Columbia
  - Howard University - IMPAACT Site, Washington D.C., District of Columbia
  - Children's Diagnostic and Treatment Center, Fort Lauderdale, Florida
  - University of Miami School of Medicine, Miami, Florida
  - University of South Florida, Tampa, Florida
  - Stroger Hospital of Cook County, Chicago, Illinois
  - Childrens Memorial Hospital, Chicago, Illinois
  - Tulane University Health Sciences Center, New Orleans, Louisiana
  - University of Maryland, Baltimore, Maryland
  - Johns Hopkins University - IMPAACT Site, Baltimore, Maryland
  - Children's Hospital of Michigan - IMPAACT Site, Detroit, Michigan
  - Mount Sinai Medical Center, Manhattan, New York
  - Montefiore Medical Center, The Bronx, New York
  - Childrens Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Jude Children's Research Center, Memphis, Tennessee
  - St. Jude Children's Research Hospital - IMPAACT Site, Memphis, Tennessee
- University of Puerto Rico, San Juan, Puerto Rico

REFERENCES:
- [Derived] Borkar SA, Yin L, Venturi GM, Shen J, Chang KF, Fischer BM, Nepal U, Raplee ID, Sleasman JW, Goodenow MM. Youth Who Control HIV on Antiretroviral Therapy Display Unique Plasma Biomarkers and Cellular Transcriptome Profiles Including DNA Repair and RNA Processing. Cells. 2025 Feb 15;14(4):285. doi: 10.3390/cells14040285. PMID 39996757
- [Derived] Kohn JN, Loop MS, Kim-Chang JJ, Garvie PA, Sleasman JW, Fischer B, Rendina HJ, Woods SP, Nichols SL, Hong S. Trajectories of Depressive Symptoms, Neurocognitive Function, and Viral Suppression With Antiretroviral Therapy Among Youth With HIV Over 36 months. J Acquir Immune Defic Syndr. 2021 Jun 1;87(2):851-859. doi: 10.1097/QAI.0000000000002653. PMID 33587499